CLINICAL TRIAL: NCT04401540
Title: Clinical and Epidemiological Characteristics of COVID-19 Infection on Babies of Prenatal COVID-19 Positive Women in Turkey
Brief Title: Characteristics of Neonatal Covid-19 in Turkey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Collaborators: Turkish Neonatal Society (Other)
Responsible Party: Principal Investigator, Mehmet Kenan Kanburoglu, Associate Professor of Pediatrics, Neonatologist, Head of Pediatrics, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: NICU-COVID-TR
Record Dates: First submitted 2020-05-22; First posted 2020-05-26 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: COVID-19; Neonatal Disease; Healthy
Keywords: Vertical Transmission
MeSH Terms: conditions — COVID-19; Infant, Newborn, Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — Nasopharyngeal, endotracheal aspirates of the neonate for Covid-19 Placenta and blood and stool samples of the neonate Milk of the mother
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aimed to investigate the clinical and epidemiological characteristics of neonates who will be born to Covid-19 positive mothers in Turkey. It is a multicentric prospective cohort study designed and destined only in Turkey. The investigators are planning to admit more than 20 Neonatal Intensive Care Units into the survey; nevertheless, the total number may change according to the prevalence of Covid-19 in neonates.

The investigators will also inquire into vertical transmission by collecting cord blood, placental, and postnatal serum samples to test for Covid-19 PCR and Covid-19 Ig M and IgG values from the neonates.

DETAILED DESCRIPTION:
The patients will be recruited by a secure database of "Trials Network" with individualized accounts. Plexus Corporation will hold data monitoring and primary analysis.

ELIGIBILITY:
Inclusion Criteria:

* Infants born to mothers with Covid-19 infection

Exclusion Criteria:

* If PCR values of mother negative, even though the clinic is preferable for Covid-19, the infant will not be recruited.

Max Age: 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The investigators will try to recruit all the babies that will be born to mothers with Covid-19 disease across Turkey.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Vertical Transmission | First 28 days of life
  Vertical transmission will be investigated by obtaining neonatal PCR samples in blood, stool and mother milk as well as Neonatal Covid-19 Ig M and Ig G values

SECONDARY OUTCOMES:
Hospital stay | First 28 days of life
  Hospital span time of the neonates in NICU
Early neonatal sepsis rate | First 3 days
  Early neonatal sepsis rate

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet K Kanburoglu, M.D., Study Director — Head of Pediatrics and Neonatology, Associate Professor
Locations (1):
- Recep Tayyip Erdogan University Medical School, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication
Access Criteria: The data will be shared in case of review requests from investigators who have an ORCHID account.

REFERENCES:
- [Result] Karimi-Zarchi M, Neamatzadeh H, Dastgheib SA, Abbasi H, Mirjalili SR, Behforouz A, Ferdosian F, Bahrami R. Vertical Transmission of Coronavirus Disease 19 (COVID-19) from Infected Pregnant Mothers to Neonates: A Review. Fetal Pediatr Pathol. 2020 Jun;39(3):246-250. doi: 10.1080/15513815.2020.1747120. Epub 2020 Apr 2. PMID 32238084
- [Result] Mimouni F, Lakshminrusimha S, Pearlman SA, Raju T, Gallagher PG, Mendlovic J. Perinatal aspects on the covid-19 pandemic: a practical resource for perinatal-neonatal specialists. J Perinatol. 2020 May;40(5):820-826. doi: 10.1038/s41372-020-0665-6. Epub 2020 Apr 10. PMID 32277162
- [Result] Liu W, Wang J, Li W, Zhou Z, Liu S, Rong Z. Clinical characteristics of 19 neonates born to mothers with COVID-19. Front Med. 2020 Apr;14(2):193-198. doi: 10.1007/s11684-020-0772-y. Epub 2020 Apr 13. PMID 32285380
- [Derived] Akin IM, Kanburoglu MK, Tayman C, Oncel MY, Imdadoglu T, Dilek M, Yaman A, Narter F, Er I, Kahveci H, Erdeve O, Koc E; Neo-Covid Study Group. Epidemiologic and clinical characteristics of neonates with late-onset COVID-19: 1-year data of Turkish Neonatal Society. Eur J Pediatr. 2022 May;181(5):1933-1942. doi: 10.1007/s00431-021-04358-8. Epub 2022 Jan 21. PMID 35061093
- [Derived] Oncel MY, Akin IM, Kanburoglu MK, Tayman C, Coskun S, Narter F, Er I, Oncan TG, Memisoglu A, Cetinkaya M, Oguz D, Erdeve O, Koc E; Neo-Covid Study Group. A multicenter study on epidemiological and clinical characteristics of 125 newborns born to women infected with COVID-19 by Turkish Neonatal Society. Eur J Pediatr. 2021 Mar;180(3):733-742. doi: 10.1007/s00431-020-03767-5. Epub 2020 Aug 10. PMID 32776309